CLINICAL TRIAL: NCT04573868
Title: National Study "AEC COVID-19" on Patients Undergoing Surgical Intervention During the SARS-CoV-2 Pandemic.
Brief Title: National Study "AEC COVID-19"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Salvador Morales Conde, Chief of the Unit of Innovation in Minimally Invesive Surgery. Associate Professor of Surgery, Hospitales Universitarios Virgen del Rocío
Other Study IDs: AEC-COVID
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Mortality
Keywords: COVID; Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently there is an important need to know the evolution, results and associated mortality of patients undergoing surgical intervention in Spain during the SARS-CoV-2 pandemic. With a national data collection, information could be obtained to guide the management of this group of complex patients operated on during the COVID-19 pandemic, with the aim of improving their treatment in the event of a second wave. The great spread of the virus and the difficulty in controlling it over time makes it a high priority for the scientific community in order to face new outbreaks.

The national study "AEC COVID-19" is a collaborative study (in the style of those carried out at European level such as Eurosurg, Globalsurg, etc.) that aims to know the evolution, results and associated mortality of patients undergoing surgical intervention in Spain during the SARS-CoV-2 pandemic. It is an observational study, with anonymized and coded data, which aims to demonstrate the following hypotheses:

* Patients with COVID-19 have high mortality.
* Patients with both oncological and benign pathologies have high morbidity.

The situation / follow-up at 7 days and 30 days after the intervention will be included in each patient.

ELIGIBILITY:
Inclusion Criteria:

Adult patients who undergo a surgical procedure during the pandemic

Exclusion Criteria:

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients who undergo a surgical procedure during the pandemic
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Patient who died after surgery 30 days after the surgical procedure

SECONDARY OUTCOMES:
Morbidity | 30 days
  Complictaions after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Morales-Conde, Principal Investigator — Asociacion Española de Cirujanos
Locations (1):
- Salvador Morales-Conde, Seville, Spain